CLINICAL TRIAL: NCT05112341
Title: Adjuvant Whole Breast Irradiation in Five Fractions Versus Fifteen Fractions in Early Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Heba Ali Elsagheer, assistant lecturer of oncolgy. sohag university hospital, Sohag University
Other Study IDs: soh-Med-21-10-17
Record Dates: First submitted 2021-10-24; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Study on Breast Cancer Patients
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1 standared hypofractonation
  Interventions: Radiation: radiation therapy
- group 2 fast forward group
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — the patient first is simulated then delineation is done

SUMMARY:
the study aiming for compairing results of hypofractionaton radiotherapy treatment in patient with early breast cancer between two arms the first arm recieving five fractions and the other arm recieving fifteen fraction

ELIGIBILITY:
Inclusion Criteria:

* age group ( 18-80) years
* breast conservation surgery
* Stages (pT1-3, pN0-1, M0) breast cancer.
* Any histological type of invasive breast cancer.
* All grades of breast cancer (I,II,III)

Exclusion Criteria:

* Stage (III or IV) breast cancer.
* Metastatic breast cancer (MBC)
* Recurrent breast cancer.
* Patients' co-morbidities that contraindicate radiotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study includes patients with early breast cancer recieving adjuvant radiotherapy in hypofractionation pattern the first arm recieving 15 fraction and the seconed arm recieving five fractions
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
1-disease free survival | 2 years
  the time free from disease
2- overall survival | 2 years
  the period time from treatment till death
3- toxicity from treatment | 2 years
  side effects from treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
adjuvant whole breast irradiation in five fractions versus fifteen fraction in early breast cancer
Supporting Information: SAP
Time Frame: 2 years

REFERENCES:
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] Mascaro A, Farina M, Gigli R, Vitelli CE, Fortunato L. Recent advances in the surgical care of breast cancer patients. World J Surg Oncol. 2010 Jan 20;8:5. doi: 10.1186/1477-7819-8-5. PMID 20089167
- [Background] Coates AS, Winer EP, Goldhirsch A, Gelber RD, Gnant M, Piccart-Gebhart M, Thurlimann B, Senn HJ; Panel Members. Tailoring therapies--improving the management of early breast cancer: St Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer 2015. Ann Oncol. 2015 Aug;26(8):1533-46. doi: 10.1093/annonc/mdv221. Epub 2015 May 4. PMID 25939896